CLINICAL TRIAL: NCT05804474
Title: A Retrospective, Multicenter, Controlled Clinical Trail: to Evaluate the Clinical Efficiency of Intracranial Aneurysm Assistive Software in the Morphological Measurement
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Wuxi No. 2 People's Hospital (Other); RenJi Hospital (Other); Shanxi Provincial People's Hospital (Other Government); Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other); Guangzhou Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Wang Shuo, Department of neurosurgery, Beijing Tiantan Hospital
Other Study IDs: QX2022-011-01
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm; Artificial Intelligence; Morphological measurement
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intracranial Aneurysms
  Interventions: Other: Observational study
- Normal Vessels
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
the goal of this clinical trail is to evaluate the clinical efficiency of intracranial aneurysm assistive software in the morphological measurement. The trail is designed as retrospective, multicenter, controlled clinical trail. Collecting probable cases images retrospectively according to inclusion criteria and exclusion criteria strictly. Controlling bias strictly, to make sure the measurement of intracranial aneurysm assistive software is evaluated reliably and precisely. In our trail, six physicions were recruited, containing three neuroradiologists, two radiologists and a residents. Software-assistant planning controls against no software-assisant planning，which aims to evaluate the improvement of morphological measurement efficiency of physicians.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75y, no gender limitation.
2. non-ruptured intracranial saccular aneurysm with specific intracranial CTA images.
3. Intracranial aneurysm was not treated.

Inclusion criteria of images:

1. the number of detector rows of Computed Tomography(CT) is more than 16 rows.
2. slice thickness ≤ 0.625mm, whole-brain image is considered.
3. Both plain scan sequences and enhancer sequence are required.

Exclusion Criteria:

1. combined with cerebral hemorrhage;
2. combined with cerevascular malformation or cerebral occupying lesion;
3. fusiform aneurysm or dissection aneurysm;
4. intracaverous internal carotid artery aneurysm;

Exclusion criteria of images:

1. none DICOM format;
2. quality score less than 3 scores;
3. metal artifacts existance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Intracranial aneurysm size | 10 years

SECONDARY OUTCOMES:
Intracranial aneurysm volume | 10 years
Intracranial aneurysm height | 10 years
Intracranial aneurysm neck diameter | 10 years
Parent artery diameter | 10 years
Intracranial aneurysm width | 10 years
Aspect ratio | 10 years
Size ratio | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China